CLINICAL TRIAL: NCT03173573
Title: A Five Part Phase 1 Study to Assess the Safety, Tolerability and Pharmacokinetic (PK) Profile of Single and Repeat Oral Doses of FDL176 in Healthy and Cystic Fibrosis (CF) Participants
Brief Title: A Study to Assess the Safety, Tolerability and PK Profile of FDL176 in Healthy and CF Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Flatley Discovery Lab LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDL176-2016-01
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: 5-part study. Part 1,3,4: parallel assignment; Part 2: cross over assignment; Part 5: single assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Part 1,3,4: Double blind; Part 2, 5: open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part 1 SAD FDL176 level 1 to 6 (Experimental): Part 1: Single dose of FDL176 test formulation Level 1 to 6 on healthy males.
  Interventions: Drug: FDL176
- Part 1 SAD Placebo (Placebo Comparator): Part 1: Single dose of Placebo for FDL176.
  Interventions: Drug: Placebo
- Part 2 SAD FDL176 at fasted state (Experimental): Part 2: single dose of FDL176 test formulation, fasted state.
  Interventions: Drug: FDL176
- Part 2 SAD FDL176 at fed state (Experimental): Part 2: single dose of FDL176 test formulation, fed state
  Interventions: Drug: FDL176
- Part 3 SAD FDL176 test formulation (Experimental): Part 3: Single dose of FDL176 test formulation on healthy females.
  Interventions: Drug: FDL176
- Part 3 SAD placebo (Placebo Comparator): Part 3: Single dose of Placebo for FDL176.
  Interventions: Drug: Placebo
- Part 4 MAD FDL176 Level 1 to 3 (Experimental): Part 4: Dose escalation of FDL176 test formulation Level 1 to 3.
  Interventions: Drug: FDL176
- Part 4 MAD Placebo (Placebo Comparator): Part 4: Dose escalation of Placebo for FDL176 Level 1 to 3.
  Interventions: Drug: Placebo
- Part 5 SAD FDL176 test formulation (Experimental): Part 5: Single dose of FDL176 test formulation.
  Interventions: Drug: FDL176

INTERVENTIONS:
Drug: FDL176 — CFTR modulator
  Arms: Part 1 SAD FDL176 level 1 to 6; Part 2 SAD FDL176 at fasted state; Part 2 SAD FDL176 at fed state; Part 3 SAD FDL176 test formulation; Part 4 MAD FDL176 Level 1 to 3; Part 5 SAD FDL176 test formulation
Drug: Placebo — Placebo for FDL176
  Arms: Part 1 SAD Placebo; Part 3 SAD placebo; Part 4 MAD Placebo

SUMMARY:
This is a 5-part study of FDL176. Part 1 is a double blind, placebo-controlled, dose escalation study in healthy male participants. Part 2 is a single dose, open-label study in healthy male participants. Part 3 is a single dose, double blind, placebo-controlled study in healthy female participants. Part 4 is a randomised, double-blind, placebo-controlled, dose-escalation study in healthy male and female participants.Part 5 is a single dose, open-label study in male and female participants with CF.

DETAILED DESCRIPTION:
This is a 5-part study. Part 1 is a double blind, placebo-controlled, dose escalation, first-in-human study to assess the safety, tolerability and PK profiles following single oral administration of FDL176 to healthy male participants. Part 2 is a single dose, open-label study in healthy male participants to determine the effect of food on the PK profile of FDL176. Part 3 is a single dose, double blind, placebo-controlled study in healthy female participants to assess the PK, safety and tolerability profiles of FDL176. Part 4 is a randomised, double-blind, placebo-controlled, dose-escalation study to assess the safety, tolerability and PK profiles following multiple oral administrations of FDL176 to healthy male and female participants. Part 5 is a single dose, open-label study in male and female participants with CF to determine the PK profile of FDL176.

ELIGIBILITY:
Inclusion Criteria (Part 1 to Part 4):

* If sexually active, must be willing to use two highly effective methods of birth control from Day 1 until 3 months after the last dose of investigational medicinal product (IMP)
* Body mass index (BMI) between 19 and 30 kg/m2 inclusive.
* Healthy as determined by the PI or delegate, based upon a medical evaluation including medical history, physical examination, laboratory tests and ECG.

Inclusion Criteria (Part 5):

* Males and females aged 18 years and older.
* Diagnosis of CF defined as a sweat chloride value ≥60 mmol/L by quantitative pilocarpine iontophoresis or two CF-causing mutations, documented in the participant's medical record.
* History of pancreatic insufficiency, documented in the participant's medical record.
* Stable CF disease as judged by the Investigator (or delegate).
* Forced expiratory volume in one second (FEV1) >40% of predicted normal for age, sex and height at screening.

Exclusion Criteria (Part 1 to 4):

* Prior or ongoing medical condition, medical history, physical findings, ECG findings or laboratory abnormality that, in the Investigator's (or delegate's) opinion, could adversely affect the safety of PK of the participant or would place the participant at increased risk.
* Surgery within the past three months prior to the first study drug administration determined by the PI or delegate to be clinically relevant.
* Alkaline phosphatase (ALP), aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN) at screening. Repeat testing at screening is acceptable for out of range values following approval by the Sponsor's Medical Monitor.
* Serum creatinine or total bilirubin > 1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
* Abnormal renal function at screening, defined as creatinine clearance <60 mL/min using the Modification of Diet in Renal Disease (MDRD) equation
* History of prolonged QT and/or QTcF interval.
* ECG with a single QTcF >450 msec in males, >460 msec in females, at Screening.
* Positive urinary drugs of abuse screen at Screening or Day -1, or positive alcohol screen at Screening or Day -1
* History of human immunodeficiency virus (HIV) or positive HIV, hepatitis B or hepatitis C results at screening.
* Use of any prescription drugs within 14 days or 5 half-lives (whichever is longer) before the first dose of IMP, unless in the opinion of the Investigator (or delegate) and the Sponsor's Medical Monitor the medication will not interfere with the study procedures or compromise participant safety. Hormonal contraceptives are allowed.
* Use of any non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days or 5 half-lives (whichever is longer) before the first dose of IMP, unless in the opinion of the Investigator (or delegate) and the Sponsor's Medical Monitor the medication will not interfere with the study procedures or compromise participant safety.
* Pregnant or nursing females. Female participants of childbearing potential must have a negative pregnancy test at the screening visit. Determination of participant eligibility will be at the discretion of the Investigator (or delegate) following consultation with the Sponsor's Medical Monitor.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, one glass (125 mL) of wine, or one (25 mL) measure of spirits.
* Current smoking or use of tobacco products or substitutes. Former smokers will be eligible, provided they have not smoked for at least 6 months before Day 1.
* Participation in another clinical trial involving receipt of an IMP within the past 90 days or exposure to more than four new chemical entities with 12 months of the first dosing day.

Exclusion Criteria (Part 5):

* A pulmonary exacerbation, or changes in therapy for pulmonary disease within 4 weeks prior to the Baseline (Day 1) visit.
* Abnormal liver function ≥3 × ULN: AST, ALT, total bilirubin.
* Serum creatinine or total bilirubin > 1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
* Abnormal renal function at screening, defined as creatinine clearance <60 mL/min using the MDRD equation.
* Hemoglobin <10 g/dL.
* History of prolonged QT and/or QTcF interval.
* ECG with a single QTcF >450 msec in males, >460 msec in females, at Screening.
* Use of ivacaftor or lumacaftor within 14 days prior to Day 1.
* Any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation, or re-initiation) in a chronic treatment/prophylaxis regimen for CF or CF related conditions within 4 weeks prior to Day 1.
* Pregnant or nursing females. Female participants of childbearing potential must have a negative pregnancy test at the screening visit. Determination of participant eligibility will be at the discretion of the Investigator (or delegate) following consultation with the Sponsor's Medical Monitor.
* Participation in another clinical trial involving receipt of an IP within the past 90 days or exposure to more than four new chemical entities with 12 months of the first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 4: Incidence of Treatment-Emergent Adverse Events. | Part 1: 4 weeks; Part 4: 6 weeks
  Part 1 and Part 4: Safety and tolerability of FDL176 in healthy male participants as determined by the incidence of adverse events (AE)s and serious adverse events(SAE)s.
Part 2, 3 and 5: Pharmacokinetic parameters, Cmax | Part 2: 5 weeks, Part 3: 4 weeks and Part 5: 4 weeks
  The pharmacokinetic parameters of FDL176: maximal plasma concentration
Part 2, 3 and 5: Pharmacokinetic parameters, Tmax | Part 2: 5 weeks, Part 3: 4 weeks and Part 5: 4 weeks
  The pharmacokinetic parameters of FDL176: maximal concentration
Part 2, 3 and 5: Pharmacokinetic parameters, AUC | Part 2: 5 weeks, Part 3: 4 weeks and Part 5: 4 weeks
  The pharmacokinetic parameters of FDL176: area under the plasma concentration curve
Part 2, 3 and 5: Pharmacokinetic parameters, CL/F | Part 2: 5 weeks, Part 3: 4 weeks and Part 5: 4 weeks
  The pharmacokinetic parameters of FDL176: clearance
Part 2, 3 and 5: Pharmacokinetic parameters, V/F | Part 2: 5 weeks, Part 3: 4 weeks and Part 5: 4 weeks
  The pharmacokinetic parameters of FDL176: apparent volume of distribution

SECONDARY OUTCOMES:
Part 2, 3, and 5: Incidence of Treatment-Emergent Adverse Events. | Part 2: 5 weeks, Part 3: 4 weeks and Part 5: 4 weeks
  Safety and tolerability of FDL176 in healthy male participants as determined by the incidence of adverse events (AE)s and serious adverse events(SAE)s.
Part 1 and 4: Pharmacokinetic parameters, Cmax | Part 1: 4 weeks; Part 4: 6 weeks
  The pharmacokinetic parameters of FDL176: maximal plasma concentration
Part 1 and 4: Pharmacokinetic parameters,Tmax | Part 1: 4 weeks; Part 4: 6 weeks
  The pharmacokinetic parameters of FDL176: maximal concentration
Part 1 and 4: Pharmacokinetic parameters,AUC | Part 1: 4 weeks; Part 4: 6 weeks
  The pharmacokinetic parameters of FDL176: area under the plasma concentration curve
Part 1 and 4: Pharmacokinetic parameters, CL/F | Part 1: 4 weeks; Part 4: 6 weeks
  The pharmacokinetic parameters of FDL176: clearance
Part 1 and 4: Pharmacokinetic parameters, V/F | Part 1: 4 weeks; Part 4: 6 weeks
  The pharmacokinetic parameters of FDL176: apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Ordonez, MD, Study Chair — Flatley Discovery Lab
Locations (3):
- Australia (3):
  - Wayne Hooper Clinic Clive Berghofer Cancer research Center, Herston, Queenland
  - Mater Hospital, South Brisbane, Queensland
  - Linear Clinical Research, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided